CLINICAL TRIAL: NCT04574635
Title: Human Papilloma Virus (HPV) Circulating Tumor DNA (ctDNA) in Cervical Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR1905; NCI-2020-06965 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ROR1905 (Other: Mayo Clinic in Rochester); 19-011924 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Infiltrating Cervical Carcinoma; Metastatic Cervical Carcinoma; Recurrent Cervical Carcinoma; Stage I Cervical Cancer FIGO 2018; Stage IA Cervical Cancer FIGO 2018; Stage IA1 Cervical Cancer FIGO 2018; Stage IA2 Cervical Cancer FIGO 2018; Stage IB Cervical Cancer FIGO 2018; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer FIGO 2018; Stage IB3 Cervical Cancer FIGO 2018; Stage II Cervical Cancer FIGO 2018; Stage IIA Cervical Cancer FIGO 2018; Stage IIA1 Cervical Cancer FIGO 2018; Stage IIA2 Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018; Stage III Cervical Cancer FIGO 2018; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IIIC Cervical Cancer FIGO 2018; Stage IIIC1 Cervical Cancer FIGO 2018; Stage IIIC2 Cervical Cancer FIGO 2018; Stage IV Cervical Cancer FIGO 2018; Stage IVA Cervical Cancer FIGO 2018; Stage IVB Cervical Cancer FIGO 2018
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Definitive chemoradiotherapy patients: Patients undergo collection of blood samples at baseline prior to the first fraction of radiation, during week 4 of radiotherapy, on the day of the final fraction of radiotherapy, at 3 months post-radiotherapy, every 3 months during years 1 and 2, and at the time of recurrence (if applicable).
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples

SUMMARY:
This study collects blood samples to determine if the DNA of HPV that causes cervical cancer can be detected in patients with cervical cancer that is new (primary), has come back (recurrent), or has spread to other places in the body (metastatic) and are undergoing treatment with surgery, radiotherapy, chemotherapy, and/or immunotherapy. Researchers may use this information to predict response (good or bad) of the cervical cancer to treatment and detect recurrent cancer sooner.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Patient has given permission to give tumor/blood sample for research testing
* Histological confirmation of adenocarcinoma, adenosquamous, or small cell carcinoma of the cervix
* Known HPV status defined as positive staining for p16 on IHC or DNA ISH for HPV
* Willingness to return to enrolling institution (Mayo Clinic Rochester or the University of Minnesota) for follow-up (during the Active Monitoring Phase of the study) or complete blood draws locally using study mail-in kits
* Consent to allow blood specimens to be shared with Mayo Clinic study personnel and potential external collaborators for sample analysis
* Definitive Chemoradiotherapy for Locally Advanced Disease (FIGO Stage IB2-IIIC)

  * FIGO 2019 Stage IB2-IIIC or not a surgical candidate
  * Plan to undergo definitive chemoradiotherapy including external beam radiotherapy, brachytherapy, and chemotherapy

Exclusion Criteria:

* Other active malignancy =< 2 years prior to registration.

  * EXCEPTIONS: Non-melanotic skin cancer
  * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for cancer
* Pregnancy or lactation
* Inability on the part of the patient to understand the informed consent to be compliant with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women ages 18 and older presenting with p16-positive or HPV-positive invasive carcinoma of the cervix cancer with plan to undergo therapy at Mayo Clinic Rochester or the University of Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with undetectable circulating tumor deoxyribonucleic acid (ctDNA) posttreatment in patients with detectable ctDNA pre-treatment | At 6 weeks post-surgery (cohort 1), at 4-6 weeks after completion of chemotherapy and radiation (cohort 2), 4-6 weeks post End of chemotherapy and radiotherapy (cohort 3), at 8 weeks after start of chemotherapy or immunotherapy (cohort 4)
  The proportion will be reported along with the exact 95% binomial confidence interval. Additionally will report the mean standard deviation and median interquartile range ctDNA post-treatment in these patients.

SECONDARY OUTCOMES:
ctDNA levels | Baseline
  Will be associated with Federation of Gynecology and Obstetrics stage and assessed using linear regression, reporting the correlation as well as the model estimates.
Clinical tumor response | At post-treatment assessment, assessed up to 2 years
  Will be assessed for association with baseline and post-treatment ctDNA using logistic regression. Depending on the number of tumor response, or non-response patients whichever is fewer, multiple variable models may be considered including additional relevant baseline covariates such as disease stage.
Radiographic tumor response | At post-treatment assessment, assessed up to 2 years
  Will be assessed for association with baseline and post-treatment ctDNA using logistic regression. Depending on the number of tumor response, or non-response patients whichever is fewer, multiple variable models may be considered including additional relevant baseline covariates such as disease stage.
Recurrence-free survival | Up to 2 years
  Baseline ctDNA and ctDNA at measured time points will be considered in Cox models.
Overall survival | Up to 2 years
  Baseline ctDNA and ctDNA at measured time points will be considered in Cox models. ctDNA other than at baseline will be considered in these models as a time dependent covariate. Depending on the number of events, multiple variable models may be considered including additional relevant baseline covariates such as disease stage.
ctDNA clearance kinetics | Up to 2 years
  Will be correlated with recurrence-free survival. ctDNA other than at baseline will be considered in these models as a time dependent covariate. Depending on the number of events, multiple variable models may be considered including additional relevant baseline covariates such as disease stage.
ctDNA conversion | Up to 2 years
  Will be correlated during the active monitoring phase with recurrence-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Allison E. Garda, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials